CLINICAL TRIAL: NCT07121517
Title: "Airway Complications in Pediatric Patients With Tracheostomies: To What Extent Can Symptoms Identified by Caregivers or Pediatricians Serve as Predictors for Airway Complications Confirmed Through Surveillance Endoscopy?"
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Ida Engqvist, Medical doctor, Principal Investigator, Karolinska Institutet
Other Study IDs: 2023-07493-01-V
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Surveillance; Endoscopy; Tracheostomy Complication; Tracheostomy Complications; Tracheostomy; Children in the Pediatric Intensive Care Unit or General Pediatric Care Unit Requiring a Central Venous Catheter
Keywords: surveillance; endoscopy; pediatric; intensive care unit; tracheostomy complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with tracheostomy undergoing at LIVA: All children under 18 years with tracheostomy undergoing follow-up through the long term intensive care unit LIVA at Karolinska University Hospital Solna, Sweden will be eligible for inclusion. This is a majority of the children living with tracheostomy in Sweden.

SUMMARY:
Study Objective:

This observational study aims to prospectively investigate to what extent tracheostomy-related complications in children are asymptomatic or associated with symptoms when detected through surveillance airway endoscopy. We also aim at investigating how reliable caregiver reports and investigations by pediatriscians are in identifying symptoms associated with severe tracheostomy-related airway complications.

Study Population:

The study population comprises children under 18 years of age undergoing follow-up at the Long-Term Intensive Care Unit (LIVA) at Karolinska University Hospital in Stockholm, Sweden.

Research Questions:

1. To what extent are tracheostomy-related complications in children asymptomatic when detected through surveillance airway endoscopy?
2. How reliable are caregiver reports in identifying symptoms associated with tracheostomy-related airway complications?

Methods:

Children scheduled for surveillance airway endoscopy are admitted to LIVA. Upon admission, the caregiver is asked to complete a short questionnaire regarding symptoms that may indicate a tracheostomy-related complication.

After the questionnaire has been completed, the child will be examined by the responsible paediatrician, with the aim of identifying any signs or symptoms that could indicate an airway complication. The examination includes physical examination and medical history conducted according to a predefined protocol.

The airway endoscopy is performed by an ENT surgeon who has not examined the patient beforehand and is not informed of the caregiver's responses nor the result of the examination by the pediatrician. However, there is no strict protocol in place to blind the surgeon to any visibly apparent symptoms or to information that may be spontaneously reported by the caregiver or paediatrician.

DETAILED DESCRIPTION:
Study Objective This observational study aims to prospectively investigate to what extent tracheostomy-related complications in children are asymptomatic or associated with symptoms when detected through surveillance airway endoscopy. We also aim at investigating how reliable caregiver reports and investigations by pediatriscians are in identifying symptoms associated with severe tracheostomy-related airway complications.

Background Children with airway obstruction due to congenital malformations, trauma, or chronic respiratory or neuromuscular conditions may require a tracheostomy. The Long-Term Intensive Care Unit (LIVA), part of the Pediatric Perioperative Medicine and Intensive Care (BPMI) at Karolinska University Hospital, has been providing specialized care for children with tracheostomies across Sweden since 1998. The care at LIVA involves assessements by a multidisciplinary team, including pediatricians, ENT specialists, pediatric anesthesiologists, nurses, physiotherapists, dietitians, speech therapists, counselors, and play therapists.

Follow-up at LIVA includes regular multidisciplinary assessments and one to two surveillance airway endoscopies under anesthesia annually, aimed at early detection of airway complications related to the tracheostomy tube. Complications such as granulomas, infections, or bleeding are often asymptomatic but can be potentially life-threatening. There is currently no national or international consensus on the optimal frequency of surveillance endoscopies, and the potential for individualizing surveillance based on risk factors, including the presentation of symptoms, remains unexplored. Given the risks associated with anesthesia, minimizing unnecessary procedures is critical.

Currently, a retrospective study is underway to examine the incidence of tracheostomy-related complications, their correlation with risk and demographic factors, and preoperative symptoms. Preliminary results indicate that 72% of patients experienced at least one tracheostomy-related complication, while only 19% exhibited symptoms prior to surveillance endoscopy according to patient records. Suprastomal granuloma was the most frequent complication observed. Interventions were required for all symptomatic patients and 71% of asymptomatic patients with identified complications. Patients using ventilators and/or cuffed cannulas had a higher incidence of complications compared to those without (88% vs. 61%, p<0.05).

Study Population The study population comprises children under 18 years of age undergoing follow-up at the Long-Term Intensive Care Unit (LIVA) at Karolinska University Hospital in Stockholm, Sweden.

Research Questions

1. To what extent are tracheostomy-related complications in children asymptomatic when detected through surveillance airway endoscopy?
2. How reliable are caregiver reports in identifying symptoms associated with tracheostomy-related airway complications?

Methods Children scheduled for surveillance airway endoscopy are admitted to LIVA. Upon admission, the caregiver is asked to complete a short questionnaire regarding symptoms that may indicate a tracheostomy-related complication.

After the questionnaire has been completed, the child will be examined by the responsible paediatrician, with the aim of identifying any signs or symptoms that could indicate an airway complication. The examination includes physical examination and medical history conducted according to a predefined protocol.

The airway endoscopy is performed by an ENT surgeon who has not examined the patient beforehand and is not informed of the caregiver's responses nor the result of the examination by the pediatrician. However, there is no strict protocol in place to blind the surgeon to any visibly apparent symptoms or to information that may be spontaneously reported by the caregiver or paediatrician.

Ethical Approval Ethical approval for the study has been obtained (Ref. No: 2023-07493-01).

ELIGIBILITY:
Inclusion Criteria:

All children, with tracheostomy, under the age of 18, undergoing scheduled surveillance airway endoscopy in anaesthesia as part of their regular follow-up at the Long term Intensive Care unit (LIVA) at Karolinska University Hospital are eligible for inclusion. Patients may be included several times during the study period.

Exclusion criteria:

All patients undergoing airway endoscopy that is not part of the surveillance airway endoscopy program will be excluded. Thus, emergency endoscopies are not included in this study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children below the age of 18 with tracheostomy undergoing follow-up through the Long term Intensive Care Unit at Karolinska University Hospital in Stockholm Sweden scheduled for surveillance airway endoscopy between sept 2025 and sept 2027. This includes the majority of children with tracheostomy in Sweden. Patients undergo airway endoscopy 1-2 times per year. One patient may be included more than one time. Estimated population size is approximately 100.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who are diagnosed with a serious tracheostomy related airway complication, without associated symptoms reported by caregiver prior to airway endoscopy. | 2 years
  Symtoms prior to surveillance endoscopy are recorded from caregiver reports and from clinical investigation by pediatrician upon admission. Airway complications detected through Surveillance Airway Endoscopy in children with Tracheostomy are recorded. Association between symptoms and identified airway complications is investigated.
Proportion of patients who are diagnosed with a serious tracheostomy related airway complication, without associated symptoms reported by a paediatrician prior to airway endoscopy. | 2 years
  Symtoms prior to surveillance endoscopy are recorded from caregiver reports and from clinical investigation by pediatrician upon admission. Airway complications detected through Surveillance Airway Endoscopy in children with Tracheostomy are recorded. Association between symptoms and identified airway complications is investigated.

SECONDARY OUTCOMES:
Proportion of patients that was diagnosed with at least one serious tracheostomy related complication during the study period. | 2 years
  Tracheostomy related complications are identified through suveillance airway endoscopy. Serious tracheostomy related complications incluce suprastomal granuloma, suprastomal prolapse, tip granuloma, tip erosion or other stoma pathology with urgent need for intervention.
Proportion of surveillance airway endoscopies identifying a serious tracheostomy related airway complication without associated symptoms reported by caregiver prior to airway endoscopy. | 2 years
  Symtoms prior to surveillance endoscopy are recorded from caregiver reports and from clinical investigation by pediatrician upon admission. Airway complications detected through Surveillance Airway Endoscopy in children with Tracheostomy are recorded. Association between symptoms and identified airway complications is investigated.
Proportion of surveillance airway endoscopies identifying a serious tracheostomy related airway complication without associated symptoms reported by pediatrician prior to airway endoscopy . | 2 years
  Symtoms prior to surveillance endoscopy are recorded from caregiver reports and from clinical investigation by pediatrician upon admission. Airway complications detected through Surveillance Airway Endoscopy in children with Tracheostomy are recorded. Association between symptoms and identified airway complications is investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Ida Engqvist, MD, Principal Investigator — LIVA, Barn PMI, Karolinska Universitetssjukhuset, Solna, Sweden
Locations (1):
- LIVA, Barn PMI, Karolinska Universitetssjukhuset Solna, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Undecided